CLINICAL TRIAL: NCT05964335
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel, 4-Arm Dose Ranging Study of the Safety and Efficacy of Nalbuphine Extended-Release Tablets (NAL ER) for the Treatment of Cough in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Cough Reduction in IPF With Nalbuphine ER
Acronym: CORAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAL03-202
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Cough; Nalbuphine
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- NAL ER 27 mg (Experimental): BID
  Interventions: Drug: NAL ER
- NAL ER 54 mg (Experimental): BID
  Interventions: Drug: NAL ER
- NAL ER 108 mg (Experimental): BID
  Interventions: Drug: NAL ER
- Placebo (Placebo Comparator): Placebo, BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAL ER — Oral tablets
  Other Names: Nalbuphine
  Arms: NAL ER 27 mg
Drug: Placebo — Oral tablets
  Arms: Placebo
Drug: NAL ER — Oral Tablets
  Other Names: Nalbuphine
  Arms: NAL ER 54 mg
Drug: NAL ER — Oral tablets
  Other Names: Nalbuphine
  Arms: NAL ER 108 mg

SUMMARY:
The main purpose of the study is to evaluate the effect of NAL ER on 24-hour cough frequency using objective digital cough monitoring and to assess safety and tolerability of NAL ER.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF as determined by the Principal Investigator based on ATS/ERS/JRS/ALAT guidelines.
* Cough Severity Score ≥ 4 on CS-NRS (Cough Severity Numerical Rating Scale) during the Screening period and Baseline.
* History of chronic cough for at least 8 weeks before screening.
* SpO2 ≥ 92%, taken after at least 5 minutes in a sitting position, undisturbed and non-stimulated (Saturation of Hemoglobin with Oxygen as Measured by Pulse Oximetry).
* FVC ≥ 40% predicted of normal - Forced Vital Capacity, as determined by spirometry adhering to ATS/ERS guidelines.
* DLCO ≥ 25% predicted of normal - Diffusing capacity of the lung for carbon monoxide corrected for hemoglobin, assessed within the last 12 weeks, or at the time of screening.

Exclusion Criteria:

* Currently on continuous oxygen therapy for longer than 16 hours at any level or delivered by any modality. Intermittent oxygen use of any duration over any given 24-hour period is allowed.
* Inadequate swallow reflex as assessed by the ability to sip 3 fluid oz (or 89 mL) of water without coughing or choking.
* Upper or lower respiratory tract infection in the last 8 weeks prior to the baseline visit.
* Clinical history of aspiration pneumonitis.
* Diagnosis of sleep apnea.
* Abnormal kidney or liver functions based on Screening lab results.
* Known hypersensitivity to nalbuphine or to NAL ER excipients
* History of major psychiatric disorder.
* History of substance abuse.
* Significant medical condition or other factors that may interfere with the participant's ability to successfully complete the study.
* Pregnant or lactating female participant.
* Known intolerance (gastrointestinal, central nervous system symptoms), hypersensitivity, drug allergy following the use of an opioid drug.
* Use of opiates is prohibited within 14 days prior to the baseline visit.
* Use of benzodiazepines are prohibited within 14 days prior to the baseline visit and for the duration of the study.
* Monoamine oxidase inhibitors (MAOIs) including methylene blue (methylthioninium chloride) and the antibiotic linezolid are prohibited within 14 days prior to the baseline visit and for the duration of the study.
* Use of oral corticosteroid cough treatment is prohibited within 4 weeks prior to the baseline visit and for the duration of the study.
* Exposure to any investigational medication, including placebo, is prohibited within 4 weeks prior to the baseline visit and for the duration of the study.
* Medications prescribed as cough suppressants are prohibited unless on a stable dose 14-days prior to the baseline visit and are expected to remain on that dose for the duration of the study.
* Use of medications that affect serotonergic neurotransmission and that when used concomitantly with opioids can increase the risk of serotonin syndrome are prohibited unless on a stable dose 14-days prior to the baseline visit and are expected to remain on that dose for the duration of the study.
* Anti-fibrotic medications are prohibited unless on a stable dose for 8 weeks prior to the baseline visit and are expected to remain on that dose for the duration of the study.
* Strong inhibitors/inducers of the P450 Isozymes are prohibited unless on a stable dose for 14-days prior to baseline visit and are expected to remain on that dose for the duration of the study.
* Use of a medication having a "known risk" of Torsade de Pointes (categorized as "KR" on the Credible Meds® website.) 4 weeks prior to Baseline.
* Use of unstable doses of medications associated with a potential risk of QT prolongation but not clearly associated with Torsade de Pointes within 4 weeks of screening.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Relative Change From Baseline in 24-hour Cough Frequency at Week 6 | Baseline, Week 6

SECONDARY OUTCOMES:
Change From Baseline in Evaluating Respiratory Symptoms in Idiopathic Pulmonary Fibrosis (E-RS:IPF) Cough subscale at Week 6 | Baseline, Week 6
Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Week 12
Relative Change From Baseline in 24-hour Cough Frequency at Weeks 2,4, and 6 | Baseline, Weeks 2, 4, and 6
Percentage of Responders With ≥30%, ≥50% and ≥75% Reduction in the 24-Hour Cough Frequency at Week 2, 4, and 6 | At Weeks 2, 4, and 6
Relative Change From Baseline in Awake Cough Frequency at Week 2, 4, and 6 | Baseline, Weeks 2, 4, and 6
Relative Change From Baseline in Sleep Cough Frequency at Week 2, 4, and 6 | Baseline, Weeks 2, 4, and 6
Change From Baseline in E-RS: IPF Cough Subscale at Weeks 1, 2, 3, 4, 5, and 6 | Baseline, Weeks 1, 2, 3, 4, 5, 6
Percentage of E-RS: IPF Cough Subscale Responders With At least one Category Improvement at Weeks 1, 2, 3, 4, 5, and 6 | At Weeks 1, 2, 3, 4, 5, and 6
Change From Baseline in E-RS: IPF Total Score, Subdomain Scores (IPF-Breathlessness, IPF-Cough, IPF-Sputum, and IPF-Chest Symptoms) and Individual Items at Weeks 1, 2, 3, 4, 5, and 6 | Baseline, Weeks 1, 2, 3, 4, 5, and 6
Change From Baseline in Cough Severity Numerical Rating Scale (CS-NRS) at Weeks 1, 2, 3, 4, 5, and 6 | Baseline, Weeks 1, 2, 3, 4, 5, and 6
Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score at Week 6 | Baseline, Week 6
Percentage of LCQ Total Score Responders With 1.3-Point Increase Response at Week 6 | At Week 6
Change From Baseline in LCQ Domains and Individual Items at Week 6 | Baseline, Week 6
Change From Baseline in Living With Pulmonary Fibrosis Impacts Questionnaire (L-IPF©) at Week 6 | Baseline, Week 6
Change From Baseline in Living With Pulmonary Fibrosis Symptoms Questionnaire (L-IPF) and its Domains at Week 6 | Baseline, Week 6
Change from Baseline in EuroQol 5-Dimension 5-Level (EQ-5D-5L™) at Week 6 | Baseline, Week 6
Change From Baseline in Patient Global Impression of Severity (PGI-S) Cough at Weeks 2, 4, and 6 | Baseline, Weeks 2, 4, and 6
Absolute Values of PGI-C Cough Score at Weeks 2, 4, and 6 | At Weeks 2, 4, and 6
Percentage of Participants With Improvement by ≥1 and ≥2 Categories, Worsening by ≥1 and ≥2 Categories, and no Change on PGI-C and PGI-S Cough at Each Post-Baseline Timepoint | At Weeks 2, 4, and 6
Change from Baseline in PGI-S IPF at Weeks 2, 4, and 6 | Baseline, Weeks 2, 4, and 6
Absolute Values of PGI-C IPF at Weeks 2, 4, and 6 | At Weeks 2, 4, and 6
Percentage of Participants With Improvement by ≥1 and ≥2 Categories, Worsening by ≥1 and ≥2 Categories, and no Change on the PGI-C and PGI-S IPF at Weeks 2, 4, and 6 | At Weeks 2, 4, and 6
Change From Baseline in Clinicians Global Impression of Severity (CGI-S) score at Week 6 | Baseline, Week 6
Absolute Values for CGI-C IPF Score at Week 6 | At Week 6
Percentage of Participants With Improvement by ≥1 and ≥2 Categories, Worsening by ≥1 and ≥2 Categories, and no Change on the CGI-C and CGI-S at Week 6 | At Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (59):
- Australia (6):
  - Eastern Health-Box Hill Hospital, Box Hill
  - Concord Repatriation General Hospital, Concord
  - Austin Hospital, Heidelberg
  - Respiratory Clinical Trials Pty Ltd, Kent Town
  - TrialsWest Pty Ltd, Spearwood
  - Westmead Hospital, Westmead
- Canada (4):
  - CIC Mauricie Inc., Trois-Rivières, Quebec
  - Dynamic Drug Advancement, Ajax
  - Centre for Lung Health Clinic, Vancouver
  - The Pacific Lung Health Centre - St. Pauls Hospital, Vancouver
- Chile (6):
  - Hospital Clinico Regional Dr. Guillermo Grant Benavente, Concepción
  - Centro de Investigaciones Medicas Cemedin Ltda., Quillota
  - Clinica Universidad de los Andes, Santiago
  - Centro de Investigacion del Maule, Talca
  - Hospital Carlos Van Buren, Valparaíso
  - Oncocentro APYS, Viña del Mar
- Germany (7):
  - Universitatsklinik Ruhrlandklinik, Westdeutsches Lungenzentrum, Essen
  - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hannover Medical School, Hanover
  - University Hospital of Leipzig, Leipzig
  - IKF Pneumologie Mainz, Helix Medical Excellence Center Mainz, Mainz
  - University Medical Center of Johannes Gutenberg-University Mainz, Mainz
  - Krankenhaus Bethanien, Solingen
- Italy (5):
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele- Ospedale Gaspare Rodolico, Catania
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Di Foggia, Foggia
  - Azienda Ospedaliera San Gerardo di Monza, Monza
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Martini Ziekenhuis, Groningen
  - Erasmus Medisch Centrum 1, Rotterdam
  - HMC (Haaglanden Medisch Centrum) Bronovo, The Hague
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego, Lodz
  - Warminsko Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Samodzielny Publiczny Wojewodzki Szpital Zespolony w Szczecinie, Szczecin
- Spain (4):
  - Clinica Mi Tres Torres Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital La Milagrosa, Madrid
  - HUMV, Santander
- Turkey (Türkiye) (6):
  - Gulhane Askeri Tip Akademisi (GATA) - Gulhane Askeri Tip Fakultesi (Gulhane Military Medical Academy and Medical School), Ankara
  - Akdeniz University Faculty of Medicine, Antalya
  - Canakkale Onsekiz Mart Universitesi (COMU) - Tip Fakultesi Hastanesi, Çanakkale
  - Sureyyapasa Gogus Hastaliklari ve Gogus Cerrahisi Egitim ve Arastirma Hastanesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Selcuk Universty Medical Faculty, Konya
- United Kingdom (13):
  - Queen Elizabeth Hospital Birmingham - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Papworth Hospital, Cambridge
  - Hull and East Yorkshire - Castle Hill Hospital, Cottingham
  - Royal Infirmary Of Edinburgh, Edinburgh
  - University College London, London
  - Royal Brompton Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Wythenshawe Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Southern Health & Social Care Trust, Craigavon Area Hospital, Portadown
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molyneaux PL, Mogulkoc N, Gunen H, Doboszynska A, Kreuter M, Neustifter B, Mathur V, Cassella J; CORAL Study Group. Oral Nalbuphine in Idiopathic Pulmonary Fibrosis-Associated Cough: The CORAL Randomized Clinical Trial. JAMA. 2026 Jan 22. doi: 10.1001/jama.2025.26179. Online ahead of print. PMID 41569557